CLINICAL TRIAL: NCT04066972
Title: Intensive Aerobic and Task-specific Training to Restore Walking and Boost Neuroplasticity Among People With MS-related Walking Disability: a Proof of Principle Trial
Brief Title: Vigorous Cool Room Treadmill Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Michelle Ploughman, Assistant Professor of Medicine, Memorial University of Newfoundland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018.088
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis; Rehabilitation; Gait Disorders, Neurologic; Neuronal Plasticity
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: This is a 'proof-of-principle/feasibility' within group repeated measures study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Other: Body-weight supported treadmill training in a room cooled to 16°C

INTERVENTIONS:
Other: Body-weight supported treadmill training in a room cooled to 16°C — A total of 30 training sessions will be conducted in 10 weeks for 30 minutes per session and 3 times per week in a cool room (16⁰ C) on a treadmill that is equipped with safety straps to prevent falls. A pneumatic harness system will be used to provide 10% body-weight support during training sessions. The participants will start exercising on the treadmill at 80% of their self-selected walking speed with 1% incline and will increase as per their tolerance (will progress weekly based on 40-65% heart rate reserve). Heart rate, perceived fatigue and rating of perceived exertion will be monitored continuously during exercise sessions. Initial training will commence with intermittent rest periods [1 to 5 minutes] as requested by the participants and will be progressed to a maximum of 30-minute continuous treadmill walking.
  Other Names: Vigorous cool room treadmill training

SUMMARY:
People with multiple sclerosis (MS) are often offered walking aids and compensatory strategies rather than restorative rehabilitation. We have developed a cool room treadmill training method that uses body-weight support that people with MS fatigue and heat sensitivity can tolerate. Our previous research shows that people with advanced MS use three times more energy for essential tasks such as walking. This project will test whether 10 weeks of body-weight supported treadmill training in a room cooled to 16°C improves walking, fitness and fatigue in people with advanced MS.

ELIGIBILITY:
Inclusion Criteria:

* clinically definite MS
* relapse-free in the previous 3 months
* requiring ambulatory assistive devices (EDSS 6.0-7.0)
* negative PAR-Q screen for risk factors
* greater than 6-weeks post Botulinum Toxin injection (if received) in the lower extremity

Exclusion Criteria:

* pregnancy or intention of becoming pregnant
* finished a drug/device study in the last 30 days
* over 75 years of age
* unable to control bowel and bladder on physical exertion
* currently attending physical rehabilitation
* having no difficulty walking in the community (self-selected walking speed >120 cm/s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting vigorous cool room treadmill training | 10 weeks
  Recruitment and retention rates
Feasibility of conducting vigorous cool room treadmill training | 10 weeks
  Incidence of adverse events
Feasibility of conducting vigorous cool room treadmill training | 10 weeks
  Degree of body-weight support provided by the harness (%)
Feasibility of conducting vigorous cool room treadmill training | 10 weeks
  Rest required (minutes)

SECONDARY OUTCOMES:
Timed 25 foot walk test | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
Spatiotemporal parameters of gait measured while walking at fast and self-selected pace | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
Fatigue severity scale | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
  A 9-item questionnaire, which assesses the severity of fatigue with items scored on a 7-point scale, '1 = strongly disagree' and '7 = strongly agree'. The minimum and maximum score possible are 9 and 63 respectively. Another reporting method is the mean of all scores from all 9-items, with minimum and maximum score possible being 1 and 7 respectively.
Modified fatigue impact scale | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
  A 21-item scale, which assesses the perceived impact of fatigue with items rated by participants on a 5-point Likert scale, '0 = never' to '4 = almost always'. The items are aggregated into total score as well as three subscales: physical, cognitive, and psychosocial. The total score ranges from 0 to 84, physical subscale from 0 to 36, cognitive subscale from 0 to 40, and psychosocial subscale from 0 to 8.
Maximal oxygen consumption during graded exercise test | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
Health-related quality of life assessed using 36-Item Short-Form Health Survey | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
Serum brain derived neurotrophic factor | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
  Resting and exercise-induced serum levels of brain derived neurotrophic factor in response to the 10-week exercise intervention
Serum interleukin-6 | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
  Resting and exercise-induced serum levels of interleukin-6 in response to the 10-week exercise intervention
Montreal cognitive assessment | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
Corticospinal excitability measured using transcranial magnetic stimulation | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
Body composition measured using dual energy x-ray absorptiometry | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
Magnetization transfer ratio measured using magnetic resonance imaging | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
Aerobic cost of walking | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
Step counts | Following completion of the 10-week exercise intervention and 3-months post-exercise intervention
  Via Accelerometry

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No
The data supporting this study are available at request from the corresponding author at the Memorial University of Newfoundland, Canada.

REFERENCES:
- [Derived] Chaves AR, Devasahayam AJ, Kelly LP, Pretty RW, Ploughman M. Exercise-Induced Brain Excitability Changes in Progressive Multiple Sclerosis: A Pilot Study. J Neurol Phys Ther. 2020 Apr;44(2):132-144. doi: 10.1097/NPT.0000000000000308. PMID 32168157
- [Derived] Devasahayam AJ, Chaves AR, Lasisi WO, Curtis ME, Wadden KP, Kelly LP, Pretty R, Chen A, Wallack EM, Newell CJ, Williams JB, Kenny H, Downer MB, McCarthy J, Moore CS, Ploughman M. Vigorous cool room treadmill training to improve walking ability in people with multiple sclerosis who use ambulatory assistive devices: a feasibility study. BMC Neurol. 2020 Jan 22;20(1):33. doi: 10.1186/s12883-020-1611-0. PMID 31969132